CLINICAL TRIAL: NCT03042195
Title: Supplementary Postoperative Parenteral Nutrition for Head and Neck Cancer Patients - A Randomized Trial
Brief Title: Supplementary Postoperative Parenteral Nutrition for Head and Neck Cancer Patients
Acronym: SpPN-HNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-16042979
Record Dates: First submitted 2016-12-08; First posted 2017-02-03 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Head and Neck Neoplasm
Keywords: Supplementary Parenteral Nutrition; Postoperative Nutrition; Postoperative complications
MeSH Terms: conditions — Head and Neck Neoplasms; Postoperative Complications | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Supplementary parenteral nutrition
  Interventions: Other: Parenteral Nutrition
- Control group (No Intervention): The control group will receive standard nutritional care

INTERVENTIONS:
Other: Parenteral Nutrition — Supplementary parenteral nutrition to achieve 100% coverage of estimated needs
  Arms: Intervention group

SUMMARY:
The purpose of the study is to examine whether postoperative nutrition with endeavours of 100% coverage of the patient's estimated energy and protein needs, can reduce the incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed head and neck cancer surgery and got a feeding tube perioperatively
* Patients of legal age
* Patients who can understand and read Scandinavian languages

Exclusion Criteria:

* Patients with allergy to components in parenteral nutrition
* Patients where it is impossible to give parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-18 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Postoperative Infectious Complications | At day 30
  Local and systemic
Postoperative Thrombotic Complications | At day 30

SECONDARY OUTCOMES:
Fistula formation without infection defined by journal documentation | Day 1,2,3,4,7,14, 23 and 30
  The measurement that will be used is documented fistula formation in the patients´ journal without increased infection parameters (c-reactive protein and leukocytes)
Number of participants who develop Refeeding Syndrome defined as a decrease in p-phosphate and clinical symptoms of refeeding syndrome; edema, dyspnea, hypertension, arrhythmia, confusion and/ or cases of spasm. | Day 2,3,4
  Data are collected from the patient's record.
Number of participants who develop Refeeding Phenomena defined as a decrease in p-phosphate without clinical symptoms of refeeding syndrome; edema, dyspnea, hypertension, arrhythmia, confusion and/ or cases of spasm. | Day 2,3,4
  Data will be collected from the patient's record.
Length of stay at the hospital | Up to 30 days
Coverage of energy requirement, estimated by the Harris Benedict formula. Coverage is estimated by daily dietary registration. | Day 1,2,3,4
Coverage of protein requirement, estimated in g/kg/day. The coverage is estimated by daily dietary registration. | Day 1,2,3, 4
Hand Grip Strength measured by a hand grip strength dynamometer in kilograms. | Baseline and Day 2,3,4

OTHER OUTCOMES:
Biochemical Changes in Liver Parameters; p-alanine aminotransferase, p-bilirubin, alkaline phosphatase and INR (international normalized ratio). | Baseline and Day 2,3,4
Number of patients who develop coagulopathy defined as increase in INR (international normalized ratio) above the reference level. | Baseline and Day 2,3,4
Presence of nausea under treatment measured by a VAS-scale (visual analogue scale). | Day 2,3,4
Presence of oedema measured by weight in kg. | Day 2,3,4
Causes of insufficient dietary intake, measured by a questionnaire filled out by the patient. | Day 2,3,4
Presence of vomiting under treatment registered by patient reported cases. | Day 2,3,4

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Ear, Nose and Throat Surgery, Rigshospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No